CLINICAL TRIAL: NCT01266954
Title: An Open Label Study To Investigate the Pharmacokinetics and Pharmacodynamics of Repeat Escalating Doses of the Oral AKT Inhibitor GSK2141795 by 18F FDG PET Analysis in Subjects With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113124
Record Dates: First submitted 2010-10-21; First posted 2010-12-24 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Solid Tumours
Keywords: Cancer; 18F FDG; PK; PET; Positron Emission Tomography; PD; AKT Inhibitor; GSK2141795
MeSH Terms: conditions — Neoplasms | interventions — GSK2141795

ARMS (2):
- Stage 1 (Experimental): Three to six patients on a medium dose of GSK2141795 for four weeks
  Interventions: Drug: GSK2141795
- Stage 2 (Experimental): Nine to eighteen subjects on a low, medium or high dose of GSK2141795 for four weeks
  Interventions: Drug: GSK2141795

INTERVENTIONS:
Drug: GSK2141795 — GSK2141795 is an oral, low nanomolar pan-AKT kinase inhibitor that demonstrates activity in hematologic and solid tumor cell lines. It also delays tumor growth in a dose dependent manner in solid tumor xenograft mouse models

SUMMARY:
The purpose of this study is to explore the potential dose response relationship between the pharmacokinetics of GSK2141795 and [18F] FDG PET pharmacodynamic markers of glucose metabolism in tumor tissue. Three to six subjects will be enrolled in each cohort and dosed with repeat escalating doses of GSK2141795. [18F] FDG PET imaging and optional tumor biopsies will be done prior to initiation of dosing and sequentially at select time points during the first five weeks of dosing. The maximal dose of a given schedule evaluated in this study will not exceed the maximal tolerated dose established in the first-time-in-human trial PCS112689 for the same schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent
2. Females of non-childbearing potential, 18 years or older with ovarian cancer
3. Histologically or cytologically confirmed diagnosis of PET-positive recurrent or persistent ovarian cancer
4. Histologically or cytologically confirmed diagnosis of PET-positive recurrent or persistent uterine or gastro-oesophageal tumors (these tumor types will only be included if there is poor enrollment of patients with ovarian cancer)
5. Disease at least 2 cm suitable for assessment by imaging
6. Performance Status score of 0, 1 or 2 according to the Eastern Cooperative Oncology Group scale
7. Adequate organ systems function

Exclusion Criteria:

1. Chemotherapy, radiotherapy, or immunotherapy within 28 days prior to the first dose of GSK2141795
2. Use of an investigational anti-cancer drug within 28 days or five half-lives, whichever is shorter, prior to the first dose of GSK2141795
3. Current use of a prohibited medication
4. Anticoagulants at therapeutic doses are permitted only after consultation with the GSK Medical Monitor
5. Presence of active gastrointestinal disease or other condition that could affect gastrointestinal absorption
6. Any major surgery within the last four weeks of screening
7. Unresolved toxicity greater than or equal to Grade 2 from previous anti-cancer therapy
8. Previously diagnosed diabetes mellitus
9. Current use of oral corticosteroids, with the exception of inhaled or topical corticosteroids
10. Any serious or unstable pre-existing medical, psychiatric, or other condition
11. Symptomatic or untreated CNS metastases or leptomeningeal involvement
12. Evidence of severe or uncontrolled systemic diseases
13. QTc interval ≥ 470 msecs
14. Other clinically significant ECG abnormalities
15. History of myocardial infarction, acute coronary syndromes
16. Class III or IV heart failure
17. Pregnant or Lactating patients
18. History of hepatitis B or C or HIV

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2011-09-01 (Actual)

PRIMARY OUTCOMES:
The amount of GSK2141795 in the blood (ng/ml) from baseline | 6 months

SECONDARY OUTCOMES:
The net unidirectional uptake of FDG (Ki) from baseline | 6 months
The change in size of tumor from baseline (RECIST Criteria) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study 113124 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113124?search=study&search_terms=113124#rs